CLINICAL TRIAL: NCT04740229
Title: Testing the Impact of Flow-based, Moderate-intensity Yoga on Executive Functioning and Stress Among Low Active Working Adults Having Symptoms of Stress
Brief Title: Moderate-intensity Flow-based Yoga Effects on Cognition and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21584
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Stress; Psychological
Keywords: sun salutations; longitudinal; remote; cognition
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity flow-based Yoga (Experimental): The intervention will consist of participants engaging in a progressive series of moderate-intensity, flow-based yoga poses, along with breathing and relaxation, for eight weeks. The intervention will be titrated in terms of supervision, with first two weeks being completely supervised, followed by partial supervision for three weeks, and three weeks of unsupervised sessions. The sessions will be ~50 minutes long, 3 times/week. All supervised sessions will be conducted online through Google Meet (GM), which is a live video interaction platform. Videos will be provided to guide unsupervised sessions. Sessions will be led by a certified yoga instructor. An orientation will be provided in the first week, given that the participants will have no or minimal experience with yoga. The intervention will consist of basic sun salutations of hatha yoga sun salutation A, sun salutation B and flow sequences, and breathing exercises, and relaxation.
  Interventions: Behavioral: Yoga
- Waitlist control (No Intervention): Participants in this group will not receive the 8-week intervention during the course of the study, and will be asked to engage in their regular activities. They will be asked to not start any new activities during the study period. After they complete the study, they will be provided with the same intervention (live instruction, feedback and supportive videos).

INTERVENTIONS:
Behavioral: Yoga — Moderate-intensity flow-based yoga movements, breathing, and relaxation for 50 minutes, 3 times per week, for 8 weeks
  Arms: Moderate-intensity flow-based Yoga

SUMMARY:
The purpose of this study is to test the efficacy of an 8-week, remotely-delivered, flow-based and moderate-intensity yoga intervention (vs. waitlist control), on stress and cognitive functioning. Participants will include individuals who are full-time working adults between the ages of 18 and 64, and currently experiencing symptoms of psychosocial stress or anxiety.

DETAILED DESCRIPTION:
Participants who pass a telephone screening, electronically sign our informed consent agreement, and complete baseline testing, will be randomized to one of two groups: yoga intervention or a waitlist control group. Before and after the 8-week intervention, participants will complete psychosocial questionnaires and computerized cognitive testing. The remote intervention will be delivered via Google Meet and will be led by a certified yoga instructor. During the course of the intervention, participants will be wearing a consumer grade accelerometer to track heart rate during yoga sessions and physical activity during the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years.
* Full-time working adults, defined as working >35 hrs/week in any industry, and not currently enrolled as a full-time student.
* Presence of at least three symptoms of stress or anxiety as measured by the symptom checklist from the Diagnostic and Statistical Manual VI.
* Low active, i.e. participating in physical activity and/or mind-body activities such as yoga and tai-chi less than 3 times/week for 30 minutes, in the last three months.
* Ability to exercise at a moderate intensity, and perform movements including sitting, standing, kicking, pulling, pushing, bending one's elbows, bending the body forward, bending one's knees, lying down and getting up without difficulty.
* No engagement in mindful activities, such as meditation, or brain training games, for greater than 3 times/week for 30 minutes, in the last three months.
* Currently not involved in any other research study or structured program related to physical activity, mind-body activities, or brain training games.
* Access to a yoga mat, and a smartphone with a data plan or access to WiFi, on which an application could be downloaded.
* Access to a laptop or desktop with an attached keyboard
* Willingness to be randomized to one of two conditions

Exclusion Criteria:

* Age below 18 years or above 64 years
* Students or non full-time working adults, such as part-time working adults
* Presence of two or less symptoms of stress or anxiety as measured by the symptom checklist from the Diagnostic and Statistical Manual VI.
* Engaging in high levels of physical activity (≥ 30 minutes, two or more times/week, for the last three months) and/or a regular practitioner of Yoga or mind-body activities such as tai-chi and mindfulness meditation (≥ 30 minutes, two or more times/week, for the last three months) and/or a certified yoga teacher.
* Mobility impairment restricting ability to engage in moderate intensity activity.
* Engagement in mindful activities, such as meditation, or brain training games, for greater than 3 times/week for 30 minutes, in the last three months
* Currently involved in research study or structured program related to physical activity, mind-body activities, or brain training games
* No access to yoga mat or a smartphone with data or WiFi, as well as refusal to download a health application on their smartphone.
* Refusal or unwillingness to be randomized into either of the conditions.
* Having any of the following medical conditions, including risk of seizure, psychiatric and/or neurological disorders, or diagnosed hypertension or blood pressure of 200/105 or more.
* Score of >1 on the Physical Activity Readiness Questionnaire.
* Unavailable for >one week in the 10-week study
* Prior yoga experience in the last 10 years. i.e. those who have engaged in 50 consecutive weeks of yoga sessions each lasting 60 minutes, without missing 12 weeks or more

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | Change from baseline at 8 weeks
  The Perceived Stress Scale (PSS), developed by Cohen, Kamarck, and Mermelstein (1983) will be used to measure perceived psychosocial stress. The PSS is a 10-item scale that measures the extent to which situations are perceived as stressful. Responses range from 0 (Never) to 4 (Very often) and higher scores indicate a higher level of perceived stress. The Brief Job Stress Questionnaire, developed by Kawada and Otsuka (2011), is a 15-item scale measuring job stress. It focuses on the evaluation of job demands, job control, job support, and degree of job satisfaction. Responses range from 1 (Agree) to 4 (Disagree) and higher scores indicate a lower level of stress.

SECONDARY OUTCOMES:
Task switching paradigm | Change from baseline at 8 weeks
  This measures cognitive flexibility, i.e. a participant's ability to adapt quickly to changing rules and the cost associated with it. In this task, participants have to characterize the picture presented according to shape or color, with a switch in the rules occurring every two tasks. Participants are cued to the rule before the stimulus is presented. Reaction time and accuracy will be recorded, with lower reaction time and higher accuracy indicating better performance. Participants will complete 40 trials.
Digit span forward and backward | Change from baseline at 8 weeks
  This is a measure of the storage and manipulation capacity of working memory. The participant will be shown a series of digits presented on PowerPoint, through screen sharing. The minimum length of digits presented is 3 (e.g., 638) and the maximum length is 9 (e.g., 628295702). In the forward task, participants will be asked to recall the digits exactly as they were presented, while in the backward task, they will have to recall them in the reverse order. Digit-span backward is the more complex task of the two. Accuracy will recorded, with higher accuracy indicating better performance.
Digit symbol substitution test (DSST) | Change from baseline at 8 weeks
  DSST is a task measuring processing speed. Participants will be shown a code-key in which every digit matches a particular symbol. Then, they will be shown a symbol on the screen and participants will have to say the corresponding digit aloud, as quickly and accurately as possible. Participants are given 90 seconds to complete as many digit-symbol pairings as possible. The number of accurate pairings will be recorded, with a higher score indicating better performance. This task will be completed by showing the symbols to participants via screen sharing.
Stroop task | Change from baseline at 8 weeks
  Stroop task measures response inhibition or response interference control. Participants will be shown a series of word colors that are either congruent or incongruent with the color of the word itself. The participant will be asked to respond to the color of the word and not the word itself. Responses are made with the keyboard. The incongruent condition is the more difficult condition of the two. Reaction time is recorded and a cost score is calculated, with shorter cost scores indicating better performance.

OTHER OUTCOMES:
Self-Compassion | Change from baseline at 8 weeks
  . Self-compassion will be assessed via the Self-Compassion Scale (Neff, 2003). It is a 26-item measure of self-compassion, with items across six subscales, namely, self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Participants answer on a Likert type response scale ranging from 1 (almost never) to 5 (almost always). A total score of general self-compassion is derived by summing all the items.
Personal optimism and self-efficacy optimism | Change from baseline at 8 weeks
  Personal optimism and self-efficacy optimism from the POSO-E (Gavrilov-Jerković, Jovanović, Žuljević, & Brdarić, 2014) will be measured. This is a 9-item scale has descriptive statements regarding optimism, and participants rate whether the statement describes them on a 4-point Likert scale, ranging from 0 (completely incorrect) to 3 (completely correct). A total score is calculated by averaging the response for each subscale, with higher scores indicating higher optimism.
Covid-related stress | Change from baseline at 8 weeks
  Participants will respond to items assessing stress caused due to the pandemic. This will include items assessing changes in their sleeping, eating habits, mental health, and work.
Self-efficacy | Change from baseline at 8 weeks
  Self-efficacy specific to yoga was assessed using the Yoga Self-efficacy Scale (Birdee, Sohl, & Wallston, 2016). It is a 12-item scale that measures self-efficacy related to engaging in yoga postures, breathing, and meditation. Responses are scored on a Likert type scale ranging from 1 (strongly disagree) to 9 (strongly agree). The response options of the scale will be modified to percentages (0% to 100%). Total score is calculated by summing all items, and a higher score reflects higher self-efficacy. Additionally, a total score was calculated separately for questions relating to postures, breathing, and meditation. Self-efficacy to engage in physical activity will be assessed using the Lifestyle Self-efficacy Scale (E McAuley et al., 2009), which asks participants about their belief in their ability to be physically active five or more times per week at a moderate intensity, for at least 30 minutes, for six months. The duration was modified to reflect the duration of the study, i.e.
Mindfulness and Attention | Change from baseline at 8 weeks
  Mindfulness will be assessed via the Mindfulness and Attention Awareness Scale (K. Brown & Ryan, 2003). It is a 15-item measure of dispositional mindfulness in the context of day to day activities. Participants answer on a Likert type response scale ranging from 1 (almost always) to 6 (almost never). The total score is calculated by summing the response to all items, and higher scores reflect a higher level of dispositional mindfulness.
Positive and Negative Affect | Change from baseline at 8 weeks
  The Positive and Negative Affect Schedule (PANAS) (Watson, Clark, & Tellegen, 1988) is a 20-item scale measuring positive and negative feeling states over the past week. Each scale has 10 adjectives describing feelings, and responses range from 1 (Very slightly or not at all) to 5 (Extremely). A total score is calculated by summing items in each subscale after reverse coding few items, and a higher score indicates higher positive or negative affect.
Experienced Bodily Changes Scale (EBCS) | Change from baseline at 8 weeks
  The EBCS (O'Connor, Rousseau, & Maki, 2004) is an 8-item scale that measures perceived physical changes such as changes in energy level, body weight, and physical appearance. Responses are scored on a 11-point Likert type scale ranging from -5 to +5, wherein 0 means 'no change,' + numbers mean improvement, and - numbers mean deterioration. Mullen (2011) found that the 8-item scale is not unidimensional and proposed a four-item version measuring physiological change, which will be used. Additionally, five questions will be added to measure changes related to other relevant dimensions such as energy level, stress, and mindfulness. These have previously been used in a dissertation study with internal reliability of .77 (J. D. Cohen, 2019).
Physical activity | Change from baseline at 8 weeks
  Physical activity at baseline will be assessed via the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GLTEQ) (Gaston Godin, 2011). The GLTEQ assesses leisure-time activity across three modes of activity: strenuous, moderate, and mild, in terms of frequency and duration. Weekly frequencies of strenuous, moderate, and mild activities were multiplied by nine, five, and three, respectively to create the total score or number of units. According to this score, 24 units or more is indicative of an active individual, whereas any score below 24 is indicative of a non-active individual.
Outcome expectations | Change from baseline at 8 weeks
  Participants' expectations about the outcomes of this intervention will be assessed using the Multidimensional Outcome Expectancies for Exercise Scale (MOEES). It is a 15-item questionnaire measuring physical outcome expectancies, social outcome expectancies, and self-evaluative outcome expectancies. Responses range from 1 (strongly disagree) to 5 (strongly agree). The total score for each subscale is calculated by summing the items, with higher scores being indicative of higher outcome expectations for exercise.
Self-regulation | Change from baseline at 8 weeks
  The Physical Activity Self-Regulation Scale (PASR-12) (Umstattd, Motl, Wilcox, Saunders, & Watford, 2009) will be used to assess the use of self-regulation strategies for engaging in physical activity. The PASR-12 is a 12-item questionnaire with responses ranging from 1 (never) to 5 (very often). A total score can be calculated by summing up responses to all the items. There are also six subscales (self-monitoring, goal-setting, social support, reinforcement, time management, and relapse prevention), however, research by our lab has found that this scale is not uni-dimensional. We will use a modified version of the scale. Higher score reflects higher use of self-regulation strategies.
Bodily pain | Change from baseline at 8 weeks
  Bodily pain will be assessed using the 2-item bodily pain subscale of Short Form-36 (Håvard Loge & Kaasa, 1998), and the Pain Visual Analogue Scale. The questions are "How much bodily pain have you had during the past 4 weeks?" with responses ranging from none to very severe, and "During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)?" with responses ranging from not at all to extremely. The total score is calculated by averaging the response to these two items, and a higher score reflects lesser pain. Pain Visual Analogue Scale is a one-item measure asking participants to rate their perceived pain in the moment, on 10-point ruler with labels of 'no pain' (0), 'moderate pain' (5) and 'worst pain' (10). Higher scores indicating a higher level of perceived pain.
Anxiety and Depression | Change from baseline at 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) is a 14-item scale measuring depression and anxiety. It includes questions such as "I feel tense or wound up" (depression) and "I feel restless as if I have to be on the move" (anxiety). Responses ranging from 0-3 on a Likert type rating scale. Total score is calculated by summing responses on seven items measuring depression, and seven items measuring anxiety. A total score of 0-7 indicates 'normal', 8-10 indicates 'borderline abnormal', and 11-21 indicates 'abnormal'. The State Trait Anxiety Inventory (STAI; (Spielberger, 2010) is a 40-item scale which measures state and trait anxiety (20 items each). Responses are scored on a Likert type scale ranging from 1 (almost never) to 4 (almost always). A total score is calculated for each subscale by summing the items (after some required reverse-coding). Higher score indicates a higher level of anxiety.
Rating of Perceived Exertion (RPE) | Change from baseline at 50 minutes (post-session)
  Participants will be asked to rate their perceived exertion after engaging in the exercise session. The modified RPE scale (Borg, 1998) is a 10-point scale ranging from 1 (no exertion at all) to 10 (maximal exertion) and it measures the perceived intensity of the exercise. It has been validated with objective measures of physical activity intensity (Day, Mcguigan, Brice, & Foster, 2004; Noble, Borg, Jacobs, Ceci, & Kaiser, 1983; Pincivero & Timmons, 2010)
Focus of Attention | Change from baseline at 50 minutes (post-session)
  Participants will be asked to rate their focus on attention via the item "During the last exercise session, where was your focus of attention?" The response range from 0 (external focus of attention) to 10 (internal focus of attention). This item has been validated (Hutchinson & Tenenbaum, 2007) and has been previously used to understand mental states in mind-body interventions (Phansikar et al., 2018)
Affect | Change from baseline at 50 minutes (post-session)
  Participants will rate their affect on the Feeling Scale (Hardy & Rejeski, 1989), ranging from 5 (very good) to -5 (very bad), with 0 meaning neutral.
Heart rate | Change from baseline at 50 minutes (post-session)
  Participants will measure their heart rate before and after the exercise session, using a freely available mobile application. Mobile applications calculate heart rate using photoplethysmography, which is the same technology used in a pulse oximeter. This technology detects fingertip pulse by using the smartphone's built-in camera to emit light and track color changes on the fingertip that are directly linked to one's pulse. Heart rate measurement using mobile applications based on photoplethysmography has been validated (Coppetti et al., 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois, Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will update these records once the data has been processed and published. We hope to do so within 1 year of data collection completion per NIH guidelines.
Access Criteria: Data will be accessible on an open site (e.g., Open Science Framework https://osf.io/) with a request to interested parties to engage with the investigative team about any publication of these data in an effort to avoid redundancy. Appropriate authorship crediting investigators involved in the parent study conceptualization, and any consultation regarding data interpretation should be sought by any researchers interested in publishing these data.

REFERENCES:
- [Derived] Phansikar M, Gothe N, Hernandez R, Lara-Cinisomo S, Mullen SP. Feasibility and impact of a remote moderate-intensity yoga intervention on stress and executive functioning in working adults: a randomized controlled trial. J Behav Med. 2023 Oct;46(5):720-731. doi: 10.1007/s10865-022-00385-4. Epub 2023 Feb 8. PMID 36754937
- See also: Full-time working adults interested in participating in the study should fill out the interest survey at this link — http://exercisetechlab.com